CLINICAL TRIAL: NCT00244205
Title: Using PCR Technology (Polymerase Chain Reaction Technology) for Monitoring Patients With Bladder Tumors - Optimizing Genanalyses for Clinical Use.
Brief Title: Identifying Methylation Biomarkers for Monitoring Bladder Tumors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Other Study IDs: Blæretumor PCR projekt
Record Dates: First submitted 2005-10-24; First posted 2005-10-26 (Estimated); Last update posted 2005-11-15 (Estimated); Status verified 2005-11

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Urination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Identifying genes methylated in urine

SUMMARY:
To investigate the methylation status of 4-6 genes in Urine and matching bladder tissue biopsies, in order to find methylation markers for use in a noninvasive test in monitoring patients with bladder tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bladder tumors and patients with benign urinary tract conditions with no clinical suspicion of bladder cancer.

Exclusion Criteria:

* Patients with competing urinary and systemic diseases, pregnant and patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Reza R Serizawa, MD, Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Copenhagen University Hospital at Herlev, Herlev, Copenhagen, Denmark